CLINICAL TRIAL: NCT05530642
Title: An Augmented Training Program for Preventing Post-Traumatic Stress Injuries Among Diverse Public Safety Personnel
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Regina (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Canadian Institute for Public Safety Research and Treatment (Unknown); Saskatchewan Ministry of Justice and Attorney General (Unknown); Association of Public Safety Communication Officials (Unknown); Frontenac Paramedic Services (Unknown); Ottawa Paramedic Service (Unknown); Paramedic Services Chiefs of Saskatchewan (Unknown); Peterborough County-City Paramedics (Unknown); Regina Fire and Protective Services (Unknown); Saskatchewan Association of Chiefs of Police (Unknown); Saskatchewan Federation of Police Officers (Unknown); Saskatchewan Health Authority - Regina Area (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2020-226
Record Dates: First submitted 2022-08-29; First posted 2022-09-07 (Actual); Last update posted 2023-12-04 (Actual); Status verified 2023-11

CONDITIONS: Posttraumatic Stress Disorder; Major Depressive Disorder; Panic Disorder; Generalized Anxiety Disorder; Trauma; Traumatic Stress Disorder; Trauma and Stressor Related Disorders; Vicarious Trauma
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Depressive Disorder, Major; Panic Disorder; Generalized Anxiety Disorder; Wounds and Injuries; Stress Disorders, Traumatic; Trauma and Stressor Related Disorders; Compassion Fatigue

STUDY DESIGN:
Intervention Model Description: The PSP PTSI Study uses a longitudinal prospective sequential experimental cohort design that engages each participant for approximately 16 months. Several practical constraints prohibited a randomized controlled trial, including resource limitations and probable interactions between PSP during and after training.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Emotional Resilience Skills Training (ERST) (Experimental): The Unified Protocol for the Transdiagnostic Treatment of Emotional Disorders (UP) is an evidence-based cognitive-behavioral intervention designed to cultivate constructive approach-oriented emotional engagement. The 13-week Emotional Resilience Training (ERST) is an adaptation of the UP designed for use as a proactive training course. The ERST frames emotional experiences as natural responses to threat, rather than pathological occurrences to avoid; as such, the ERST is well-suited for mitigating health challenges and the skills may also help PSP to support persons in distress, including other PSP and the community members they all serve. The ERST training materials include an instructor guide, didactic PowerPoints, and a trainee workbook.
  Interventions: Behavioral: Emotional Resilience Skills Training (ERST)

INTERVENTIONS:
Behavioral: Emotional Resilience Skills Training (ERST) — The ERST training is designed as a "train the trainer" model. Sauer-Zavala, a co-developer of the UP, personally trained a group of PSP trainers from each of the PSP pilot sectors (i.e., CanOps, Regina Fire & Protective Services, Regina Police Service, Saskatoon Police Service, Regina Emergency Medical Services, Ottawa Emergency Medical Services) during a week-long interactive workshop. The trainers continue to have access to Sauer-Zavala for optional follow-up consultation and support related to delivery of the ERST training for questions or to address any issues that arise during training. Having consultation and support available for the trainers should help to offset concerns raised about ensuring training fidelity subsequent to other mental health programs. Participants have ongoing access to ERST to support skill retention after training is completed, which should help to offset previous indications of problems with skill development for mental health programs.
  Other Names: The Unified Protocol for the Transdiagnostic Treatment of Emotional Disorders (UP)

SUMMARY:
Public safety personnel (PSP; e.g., border services personnel, correctional workers, firefighters, paramedics, police, public safety communicators) are frequently exposed to potentially psychologically traumatic events. Such events contribute to substantial and growing challenges from posttraumatic stress injuries (PTSIs), including but not limited to posttraumatic stress disorder. The PSP PTSI Study has been designed to evaluate an evidence-informed, proactive system of mental health assessment and training among Royal Canadian Mounted Police (www.rcmpstudy.ca) for delivery among diverse PSP (i.e., firefighters, municipal police, paramedics, public safety communicators). The training is based on the Unified Protocol for the Transdiagnostic Treatment of Emotional Disorders, adapted for PSP, and named Emotional Resilience Skills Training (ERST). The subsequent PSP PTSI Study results are expected to benefit the mental health of all participants and, ultimately, all PSP.

DETAILED DESCRIPTION:
Public safety personnel (PSP; e.g., border services personnel, correctional workers, firefighters, paramedics, police, public safety communicators) are frequently exposed to potentially psychologically traumatic events. Such events contribute to substantial and growing challenges from posttraumatic stress injuries (PTSIs), including but not limited to posttraumatic stress disorder. The PSP PTSI Study has been designed to evaluate an evidence-informed, proactive system of mental health assessment and training among Royal Canadian Mounted Police (www.rcmpstudy.ca) for delivery among diverse PSP (i.e., firefighters, municipal police, paramedics, public safety communicators). The training is based on the Unified Protocol for the Transdiagnostic Treatment of Emotional Disorders, adapted for PSP, and named Emotional Resilience Skills Training (ERST). Specifically, the PSP PTSI Study will: 1) adapt, implement, and assess the impact of a system for ongoing (i.e., annual, monthly, daily) evidence-based assessments; 2) evaluate associations between demographic variables and PTSI; 3) longitudinally assess individual differences associated with PTSI; and, 4) assess the impact of providing diverse PSP with a tailored version of the ERST originally developed for the Royal Canadian Mounted Police in mitigating PTSIs based on the Unified Protocol for the Transdiagnostic Treatment of Emotional Disorders. Participants are assessed at pre-training; week 1 (i.e., Time 1) and post-training; week 13 (i.e., Time 2), and then at a 1-year follow-up after training, during week 65 (Time 3). The assessments include clinical interviews, self-report surveys including brief daily and monthly assessments, and daily biometric data. The PSP PTSI Study hypotheses were pre-registered with aspredicted.org for the PSP PTSI Study and associated hypotheses occurred on March 7, 2022 with the name, "An Augmented Training Program for Preventing Post-Traumatic Stress Injuries Among Diverse Public Safety Personnel" (#90136). Hypotheses specific to individual difference variables are publicly available; however, the overarching PSP PTSI Study hypotheses are: 1) participant mental health disorder prevalence at Time 1, based on Clinical Interviews or screening tools based on self-reported symptoms, will be higher than would be expected for the general population; 2) from Time 1 to Time 2, participants will evidence reductions in risk, increases in resiliency, and improvements in mental health, as a function of the ERST; 3) participants will evidence statistically significant predictive relationships between completing assessments and changes to individual differences over time (i.e., inversely with risk, positively with resilience, positively with mental health); 4) participants will evidence statistically significant sequential predictive relationships for environmental factors or individual differences reported during the Daily Assessments, Monthly Assessments, and Full Assessments; 5) all participants will evidence sustained reductions in risk, increases in resilience, and increases in mental health at Time 3 relative to Time 2; 6) participants will evidence a statistically significant relationship between changes in individual differences over time and engagement with ERST content; 7) participants will evidence a statistically significant relationship between changes in environmental factors or individual differences over time, frequency of exercise, and other self-reported indicators of physical health; 8) relative to men, women will report more difficulties with mental disorder symptoms and occupational stressors; 9) diastole will be reduced in PSP who report symptoms consistent with one or more PTSI; 10) the biometric data will be statistically significantly and substantively correlated with measures of PTSI; 11) there will be a statistically significant and substantive relationship between PTSI symptom severity and reduced diastolic function; and 12) changes in biological variables (i.e., autonomic nervous system reactivity, heart rate variability, cardiac mechanical changes) will be associated with environmental factors or individual differences. The subsequent PSP PTSI Study results are expected to benefit the mental health of all participants and, ultimately, all PSP.

ELIGIBILITY:
Inclusion Criteria:

* Currently serving PSP firefighters, municipal police officers, paramedics, and public safety communicators
* Potential participants were Canadian citizens or permanent residents
* 18 years or older
* Fluently read, write, and speak either English or French
* Employed in their PSP sector for a minimum of three years
* Access to a computer with internet service

Exclusion Criteria:

* High risk of suicide or previous suicide attempt/hospitalization within the prior year
* Currently experiencing psychosis, mania
* Currently experiencing impairing drug or alcohol addictions
* Current or ongoing performance management concerns
* Any history of advocating against mental health care

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 192 (Actual)
Dates: Start 2020-09-22 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Posttraumatic Stress Disorder Symptoms from Time 1 (pre-training; week 1) to Time 2 (post-training; week 13) | Time 1 (pre-training; week 1), Time 2 (post-training; week 13)
  Posttraumatic Stress Disorder Checklist Version 5; Total scores range from 0 to 80; Higher scores indicate more severe symptoms.
Sustained Posttraumatic Stress Disorder Symptoms from Time 2 (post-training; week 13) to Time 3 (1-year follow-up; week 65) | Time 2 (post-training; week 13), Time 3 (1-year follow-up; week 65)
  Posttraumatic Stress Disorder Checklist Version 5; Total scores range from 0 to 80; Higher scores indicate more severe symptoms.
Change in Major Depressive Disorder Symptoms from Time 1 (pre-training; week 1) to Time 2 (post-training; week 13) | Time 1 (pre-training; week 1), Time 2 (post-training; week 13)
  Patient Health Questionnaire - 9 (PHQ-9); Total scores range from 0 to 36; Higher scores indicate more severe symptoms.
Sustained Major Depressive Disorder Symptoms from Time 2 (post-training; week 13) to Time 3 (1-year follow-up; week 65) | Time 2 (post-training; week 13), Time 3 (1-year follow-up; week 65)
  Patient Health Questionnaire - 9 (PHQ-9); Total scores range from 0 to 36; Higher scores indicate more severe symptoms.
Change in Generalized Anxiety Disorder Symptoms from Time 1 (pre-training; week 1) to Time 2 (post-training; week 13) | Time 1 (pre-training; week 1), Time 2 (post-training; week 13)
  Generalized Anxiety Disorder Scale - 7 (GAD-7); Total scores range from 0 to 28; Higher scores indicate more severe symptoms.
Sustained Generalized Anxiety Disorder Symptoms from Time 2 (post-training; week 13) to Time 3 (1-year follow-up; week 65) | Time 2 (post-training; week 13), Time 3 (1-year follow-up; week 65)
  Generalized Anxiety Disorder Scale - 7 (GAD-7); Total scores range from 0 to 28; Higher scores indicate more severe symptoms.
Change in Panic Disorder Symptoms from Time 1 (pre-training; week 1) to Time 2 (post-training; week 13) | Time 1 (pre-training; week 1), Time 2 (post-training; week 13)
  Panic Disorder Severity Scale (PDSS); Total scores range from 0 to 28; Higher scores indicate more severe symptoms.
Sustained Panic Disorder Symptoms from Time 2 (post-training; week 13) to Time 3 (1-year follow-up; week 65) | Time 2 (post-training; week 13), Time 3 (1-year follow-up; week 65)
  Panic Disorder Severity Scale (PDSS); Total scores range from 0 to 28; Higher scores indicate more severe symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: R. Nicholas Carleton, PhD, Principal Investigator — University of Regina
Locations (1):
- University of Regina, Regina, Saskatchewan, Canada

IPD SHARING:
Plan to Share IPD: No
There are ethical and privacy concerns with respect to sharing the participant data, even after anonymization; as such, requests to access the datasets should be directed to the primary investigator and will be addressed on a case-by-case basis in connection with the University of Regina Research Ethics Board.

REFERENCES:
- [Background] Carleton RN, Kratzig GP, Sauer-Zavala S, Neary JP, Lix LM, Fletcher AJ, Afifi TO, Brunet A, Martin R, Hamelin KS, Teckchandani TA, Jamshidi L, Maguire KQ, Gerhard D, McCarron M, Hoeber O, Jones NA, Stewart SH, Keane TM, Sareen J, Dobson K, Asmundson GJG. The Royal Canadian Mounted Police (RCMP) Study: protocol for a prospective investigation of mental health risk and resilience factors. Health Promot Chronic Dis Prev Can. 2022 Aug;42(8):319-333. doi: 10.24095/hpcdp.42.8.02. PMID 35993603
- [Derived] Nisbet J, Maguire KQ, Teckchandani TA, Shields RE, Andrews KL, Afifi TO, Brunet A, Keane TM, Kratzig GP, MacPhee RS, Martin RR, McCarron MCE, Neary JP, Sauer-Zavala S, Carleton RN. Suicidal Ideation, Planning, and Attempts Changes Among Diverse Canadian Public Safety Personnel After the Emotional Resilience Skills Training. Suicide Life Threat Behav. 2025 Feb;55(1):e13168. doi: 10.1111/sltb.13168. PMID 39927828
- [Derived] Carleton RN, Sauer-Zavala S, Teckchandani TA, Maguire KQ, Jamshidi L, Shields RE, Afifi TO, Nisbet J, Andrews KL, Stewart SH, Fletcher AJ, Martin R, MacPhee RS, MacDermid JC, Keane TM, Brunet A, McCarron M, Lix LM, Jones NA, Kratzig GP, Neary JP, Anderson G, Ricciardelli R, Cramm H, Sareen J, Asmundson GJG. Mental health disorder symptom changes among public safety personnel after emotional resilience skills training. Compr Psychiatry. 2025 Apr;138:152580. doi: 10.1016/j.comppsych.2025.152580. Epub 2025 Feb 5. PMID 39923735
- [Derived] Carleton RN, McCarron M, Kratzig GP, Sauer-Zavala S, Neary JP, Lix LM, Fletcher AJ, Camp RD 2nd, Shields RE, Jamshidi L, Nisbet J, Maguire KQ, MacPhee RS, Afifi TO, Jones NA, Martin RR, Sareen J, Brunet A, Beshai S, Anderson GS, Cramm H, MacDermid JC, Ricciardelli R, Rabbani R, Teckchandani TA, Asmundson GJG. Assessing the impact of the Royal Canadian Mounted Police (RCMP) protocol and Emotional Resilience Skills Training (ERST) among diverse public safety personnel. BMC Psychol. 2022 Dec 9;10(1):295. doi: 10.1186/s40359-022-00989-0. PMID 36494748
- See also: PSP PTSI Study Website — https://www.saskptsistudy.ca
- See also: RCMP Study Website — https://www.rcmpstudy.ca